CLINICAL TRIAL: NCT02160860
Title: Epidemiology of Helicobacter Pylori Infection Among Shanghai Children
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Principal Investigator, Ying HUANG, Director of Gastroenterology of Children's Hospital of Fudan University, Children's Hospital of Fudan University
Other Study IDs: HY201405-HP
Record Dates: First submitted 2014-06-04; First posted 2014-06-11 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2016-08

CONDITIONS: Bacterial Infection Due to Helicobacter Pylori (H. Pylori)

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — serum will be storage in to -80℃ fridge for further test. other biospecimen will be test at site and disposed.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Children: Children

SUMMARY:
Epidemiology of Helicobacter Pylori Infection Among Shanghai Children.

DETAILED DESCRIPTION:
To get an understanding of the Hp infection general situation and provide evidence for Hp control, we are planning to run a free physical examination and lab test for a group of children. We are going to proceed with Hp-IgG test, 13C urea breath test and salivary Hp urea antigen test together to screening and diagnosing it.

ELIGIBILITY:
Inclusion Criteria:

* Age 3~18
* Not been Clinical diagnosis of

Exclusion Criteria:

* Had antibiotics in the past week
* Had Bismuth or PPI

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Age 3~18 children
Sampling Method: Non-Probability Sample
Enrollment: 1997 (Actual)
Dates: Start 2014-05; Primary Completion 2015-09 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
HP Infection Rate Estimation for Shanghai Children | Sampling complete before June 30, 2014. Lab test finish within 10 weeks. Report release within 3 weeks after all test finished.
  Get the population of infection with HP and calculate the infection rate for the sampling group, to estimate the infection rate for whole population of Shanghai children

CONTACTS AND LOCATIONS:
Overall Officials: HAUNG Ying, Doctor, Study Director — Director of GI Department of Children's Hospital of Fudan University
Locations (1):
- Pujiang Community Health Service Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No